CLINICAL TRIAL: NCT01032876
Title: Randomized Controlled Trial on Deep Hypothermic Circulatory Arrest Versus Antegrade Cerebral Perfusion During Neonatal Cardiac Surgery
Brief Title: Cerebral Perfusion During Neonatal Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Prof. F. Haas, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08-090/K
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Congenital Heart Defects; Hypoplastic Left Heart Syndrome; Aortic Coarctation
Keywords: Congenital Heart disease; Cardiopulmonary bypass; Neonatal brain injury; Deep Hypothermic Circulatory Arrest; Antegrade Cerebral Perfusion
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome; Aortic Coarctation | interventions — Circulatory Arrest, Deep Hypothermia Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep Hypothermic Circulatory Arrest (Experimental)
  Interventions: Procedure: Deep Hypothermic Circulatory Arrest
- Antegrade Cerebral Perfusion (Experimental)
  Interventions: Procedure: Antegrade Cerebral Perfusion

INTERVENTIONS:
Procedure: Deep Hypothermic Circulatory Arrest — DHCA will be employed for a maximum of 60 minutes. If more time (>60 min) is needed for the arch reconstruction the surgeon will proceed with ACP, which will be continued for the rest of the operation (= DHCA+ACP).
  Arms: Deep Hypothermic Circulatory Arrest
Procedure: Antegrade Cerebral Perfusion — One cannula will be advanced into the brachiocephalic/ innominate artery via the usual arterial cannulation site in the aorta ascendens. A flow of 20-25% of the maximum CPB-flow will be used, which corresponds to a flow rate of 40-50 ml/ kg/ min.
  Arms: Antegrade Cerebral Perfusion

SUMMARY:
Neonates with a congenital heart defect are often in need of early cardiac surgery. In complex congenital heart defects, cardiopulmonary bypass is usually employed, with or without deep hypothermic circulatory arrest (DHCA). The brain is especially vulnerable to ischemic injury, which puts neonates undergoing complex operations at high risk of neurodevelopmental disorders. Selective antegrade cerebral perfusion (ACP) instead of DHCA during these complex operations may contribute to less cerebral damage, but literature is not conclusive on this issue.

Therefore, the investigators will perform a randomised controlled trial comparing DHCA and ACP in neonatal aortic arch reconstructions, focusing on cerebral damage and neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* Aortic arch reconstruction (diagnosis of hypoplastic left heart syndrome, hypoplastic aortic arch, severe coarctation and/ or interrupted aortic arch)
* Infants <4 months old

Exclusion Criteria:

* Anticipated arch reconstruction time longer than 60 minutes
* Sedation and intubation especially for the pre-operative MRI-scan of this research project
* Participation in another clinical trial
* Failure of data collection

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
New or worsened lesions on postoperative MRI-scan (as compared to pre-operative scan). | Approximately 1 week postoperatively

SECONDARY OUTCOMES:
Mortality within 30 days | 30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Felix Haas, MD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Algra SO, Jansen NJ, van der Tweel I, Schouten AN, Groenendaal F, Toet M, van Oeveren W, van Haastert IC, Schoof PH, de Vries LS, Haas F. Neurological injury after neonatal cardiac surgery: a randomized, controlled trial of 2 perfusion techniques. Circulation. 2014 Jan 14;129(2):224-33. doi: 10.1161/CIRCULATIONAHA.113.003312. Epub 2013 Oct 20. PMID 24141323
- [Derived] Algra SO, Groeneveld KM, Schadenberg AW, Haas F, Evens FC, Meerding J, Koenderman L, Jansen NJ, Prakken BJ. Cerebral ischemia initiates an immediate innate immune response in neonates during cardiac surgery. J Neuroinflammation. 2013 Feb 7;10:24. doi: 10.1186/1742-2094-10-24. PMID 23390999
- [Derived] Algra SO, Schouten AN, van Oeveren W, van der Tweel I, Schoof PH, Jansen NJ, Haas F. Low-flow antegrade cerebral perfusion attenuates early renal and intestinal injury during neonatal aortic arch reconstruction. J Thorac Cardiovasc Surg. 2012 Dec;144(6):1323-8, 1328.e1-2. doi: 10.1016/j.jtcvs.2012.03.008. Epub 2012 Apr 13. PMID 22503201